CLINICAL TRIAL: NCT04375020
Title: GABA From Medical Nutrition to Pancreatic Beta-cell Regeneration
Brief Title: GABA and Beta-cell Regeneration
Status: Completed | Type: Observational
Sponsor: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Principal Investigator, mahmoud younis, consultant, Ministry of Health and Population, Egypt
Other Study IDs: icel
Record Dates: First submitted 2020-05-02; First posted 2020-05-05 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1diabetes, gaba
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group1 on GABA: The first group was on insulin therapy in the form of toujeo once daily and Novorapid 3 times daily and they received GABA nutritional supplement 750mg per day.
  Interventions: Drug: GABA
- group 2 on just insulin: The second group was only on insulin injection in the form of toujeo once daily and Novorapid 3 times daily.

INTERVENTIONS:
Drug: GABA — GABA nutritional supplement 750mg per day for 6 months
  Groups: group1 on GABA

SUMMARY:
GABA(gamma-Aminobutyric acid) may be used for decreasing anti-gad antibodies and leads beta-cell regeneration.

DETAILED DESCRIPTION:
100 patients with type I diabetes were in 2 groups, had been monitored in a private clinic, number 50 each group, with 30 females and 20 males after the written consent of all patients.

All the patients Lied between 18-25 years old with 5-10 years of diabetes onset.

The first group was on insulin therapy in the form of toujeo once daily and Novorapid 3 times daily and they received GABA nutritional supplement 750mg per day.

The second group was only on insulin injection in the form of toujeo once daily and Novorapid 3 times daily.

In the first group;the investigator measured fasting c peptide levels before and after 6 months of GABA 750mg daily.Also,the investigator measured anti gad antibodies before and after 6 months of treatment.

In the second group,the investigator measured c peptide levels and anti-gad antibodies at the beginning of the trial and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

- type 1 diabetes patients age from 18 to 25 years on basal bolus insulin

Exclusion Criteria:

thyroid problems liver disease kidney disease

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: observation prospective study 100 patients with type I diabetes were int 2 groups, had been monitored in a private clinic, number 50 each group, with 30 females and 20 males after the written consent of all patients.
  All the patients Lied between 18-25 years old with 5-10 years of diabetes onset.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
gaba decrease anti gad antibodies | 6 months
  gaba 750 mg daily for type 1 diabetes patients
gaba improve c peptide levels | 6 months
  gaba 750 mg pe day for type 1 diabetes patients

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud Younis, Cairo, Egypt